CLINICAL TRIAL: NCT05732233
Title: Randomized Clinical Trial of the Ultivision AI Artificial Intelligence System for Colorectal Cancer Screening or Surveillance in Colonoscopy
Brief Title: RITUAL Ultivision AI CADe Randomized Controlled Trial
Acronym: RITUAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to discontinue the study. Discontinuation is not related to any patient safety or performance issues.
Sponsor: Satisfai Health, Inc. (Industry)
Collaborators: Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STF-2023-01
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-02

CONDITIONS: Colon Adenoma; Polyp of Colon; Adenoma Colon
Keywords: Screening; Surveillance; Artificial Intelligence; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Parallel trial design
Who Masked: Outcomes Assessor
Masking Description: Pathologist is blind to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ultivision AI colonoscopy (CADe Arm) (Experimental): Ultivision AI is used to aid in real-time detection of adenomas.
  Interventions: Device: Ultivision AI
- Standard colonoscopy (Control Arm) (Active Comparator): Patients will undergo standard colonoscopy without AI.
  Interventions: Device: Ultivision AI

INTERVENTIONS:
Device: Ultivision AI — Ultivision AI is a computer-assisted detection (CADe) device intended to aid endoscopists in the real-time identification of colonic mucosal lesions (such as polyps and adenomas) in adult patients undergoing colorectal cancer screening and surveillance examinations.

SUMMARY:
Ultivision AI is a computer-assisted detection (CADe) device intended to aid endoscopists in the real-time identification of colonic mucosal lesions (such as polyps and adenomas).

Ultivision AI CADe is indicated for white light colonoscopy only.

DETAILED DESCRIPTION:
Ultivision AI contains an image processing software and algorithm based on machine learning technology and convolutional neural networks (CNN).

The algorithm's primary function is to identify and highlight the likelihood of the presence of a colon polyp.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 to 75 years;
2. Screening or surveillance colonoscopy.
3. Iinformed consent

Exclusion Criteria:

1. Colorectal cancer;
2. Inflammatory bowel disease, including Crohn's disease or ulcerative colitis;
3. Polyposis syndrome including Familial Adenomatous Polyposis, Cowden syndome, Linch syndrome, Peutz-Jeghers syndrome, MUITYH associated polyposis, familial Colorectal Cancer type X;
4. Positive Fecal Immunochemical Test;
5. Use anti-platelet agents or anticoagulants that prevent polyps removal;
6. Colon resection, not including the appendix;
7. Subject is pregnant or lactating.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Adenoma per Colonoscopy (APC) | During the procedure/surgery
  Superiority of Ultivision-AI arm versus control arm. APC is defined as the total number of histologically confirmed adenomas resected divided by the total number of colonoscopies.
Adenoma Per Extraction (APE). | During the procedure/surgery
  Non inferiority of Ultivision-AI arm versus control arm. Where APE is the fraction of adenoma, sessile serrated lesions, and large (>10mm) hyperplastic polyps of the proximal colon (caecum, ascending colon, hepatic flexure, and transverse colon) out of total number of resections.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - UC Irvine, Irvine, California
  - University of Kansas Medical Center, Kansas City, Kansas
- University of Montreal Research Center (CRCHUM), Montréal (Québec), Montreal, Canada
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Urban G, Tripathi P, Alkayali T, Mittal M, Jalali F, Karnes W, Baldi P. Deep Learning Localizes and Identifies Polyps in Real Time With 96% Accuracy in Screening Colonoscopy. Gastroenterology. 2018 Oct;155(4):1069-1078.e8. doi: 10.1053/j.gastro.2018.06.037. Epub 2018 Jun 18. PMID 29928897
- See also: Satisfai Health — https://satisfai.health/
- See also: Meditrial Clinical Research Organization — https://www.meditrial.net/